CLINICAL TRIAL: NCT02909244
Title: Study of Gut Microbiota in Primary Immune Deficiencies, Possibly Associated With Inflammatory Bowel Disease (Chronic Granulomatous Disease, XIAP Gene Deficiency, or TTC7A Gene Deficiency)
Brief Title: Study of Gut Microbiota in Primary Immune Deficiency, Possibly Associated With Inflammatory Bowel Disease
Acronym: DIPobiota
Status: Completed | Type: Observational
Sponsor: Imagine Institute (Other)
Collaborators: Saint Antoine University Hospital (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: IMIS2014-02
Record Dates: First submitted 2016-09-05; First posted 2016-09-21 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Primary Immune Deficiencies
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Feces samples collected on all patients for study of gut microbiota
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with PID: Biological sampling: collection of feces. In case of blood samples availability in hospital biobank : analyzes of these samples in the frame of this research
  Interventions: Biological: Biological sampling
- Control patients, with no PID: Biological sampling: collection of feces.
  Interventions: Biological: Biological sampling

INTERVENTIONS:
Biological: Biological sampling — Biological sampling

SUMMARY:
Some Primary Immune Deficiencies can be associated with an inflammatory bowel disease, mimicking Crohn disease : the Chronic Granulomatous Disease (CGD), the XIAP deficiency, and the TTC7A deficiency.

This inflammatory bowel disease is frequent but inconstant, raising questions about other factors contributing to the disease. The aim of our study is to analyze, describe and compare the gut microbiota of patients with those primary immune deficiency, with or without intestinal disease.

The investigators can expect, in the long term, to compare on a same patient, the gut microbiota evolution, and to assess the role of gut microbiota modifications on the onset of an inflammatory bowel disease.

DETAILED DESCRIPTION:
The investigators will include patients (adults or children), with Primary Immune Deficiency (CGD, XIAP or TTC7A deficiencies), and they will collect feces samples from them.

In parallel, as control groups, patients with no inflammatory bowel disease and no primary immune deficiency will be included, and also patients suffering from Crohn's disease without known primary immune deficiency.

The laboratory collaborators will then realize analyzes on the microbiota collected for all patients.

The study team will then analyze the microbiota composition of the different types of patients, and try to identify some factors, associated with the appearance of an inflammatory disease on these patients.

ELIGIBILITY:
Inclusion Criteria (Patients with one of the 3 specific PID mentioned above):

* Presenting a Primary Immune Deficiency (CGD, XIAP ou TTC7A deficiency) with or without inflammatory digestive disease

Inclusion Criteria (Control patients without one of the 3 specific PID mentioned above):

* No antibiotic treatment in the month preceding the inclusion

Exclusion Criteria (all patients):

* Patients having a received a gene therapy or a Hematopoietic stem cell transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion of patients with PID Inclusion of control patients, without PID
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of factors associated with the onset of an inflammatory colitis in patients with three Primary Immuno-Deficiencies, identified in the study population | 3 years and 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Latour, Study Director — Imagine Institute; Alain Fischer, Study Chair — Imagine Institute; Harry Sokol, Study Chair — Saint-Antoine Hospital; Olivier Join-Lambert, Study Chair — Necker - Enfants malades Hospital
Locations (3):
- France (3):
  - CHRU, Lille
  - Saint-Louis Hospital, Paris
  - Necker - Enfants Malades Hospital, Paris

IPD SHARING:
Plan to Share IPD: No